CLINICAL TRIAL: NCT00192816
Title: Pain Perception in Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: 2038CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2005-09

CONDITIONS: Dementia Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: reaction to pain

SUMMARY:
The purpose of this study is to determine response to pain in Alzheimer's disease.We plan to study the effect of diffuse noxious inhibitory controls(counterirritation phenomenon)and the autonomic nervous system reaction(reflected by the heart rate) in Alzheimer's disease. The study's hypothesis is that pain perception and autonomic nervous system reaction are altered in Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

- Clinical diagnosis of Alzheimer's disease Must be able to understand a simple pain scale

Exclusion Criteria:

Neuropathy Psychotropic drugs use -

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aharon-Peretz, Study Director — Rambam Health Care Campus
Locations (1):
- Neurocognitive unit,Neurophysiology laborator Rambam Health Care Campus, Haifa, Israel